CLINICAL TRIAL: NCT07251166
Title: A Multi-center, Open-label, Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumor Efficacy of GenSci140 in Patients With Advanced Solid Tumors
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of GenSci140 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GenSci140-101
Record Dates: First submitted 2025-11-14; First posted 2025-11-26 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Level 1~ Dose Level 5 (Experimental): Participants who meet the inclusion criteria and do not meet the exclusion criteria will be sequentially enrolled into five pre-specified doses for dose groups 1-5.
  Interventions: Drug: GenSci140 for Injection
- Cohort 1~ Cohort 4 (Experimental): Cohort 1: Cohort 1 is planned to be conducted in patients with ovarian cancer. Cohort 2: FRα-positive endometrial cancer. Cohort 3: FRα-positive lung cancer. Cohort 4: FRα-positive triple negative breast cancer.
  Interventions: Drug: GenSci140 for Injection

INTERVENTIONS:
Drug: GenSci140 for Injection — Participants will receive GenSci140 on Day 1 of each 21-day cycle. GenSci140 will be administered until unacceptable toxicity, disease progression, withdrawal of informed consent, death, loss to follow-up, or initiation of new anti-tumor therapy (whichever occurs first).

SUMMARY:
This is a phase I, multi-center, open-label, dose-escalation (Part 1) and dose-expansion (Part 2) first-in-human study in China to evaluate the safety, tolerability, PK profile and efficacy of GenSci140 in participants with advanced solid tumors, and to determine the MTD (if any) and RDE. The dose-expansion study aims to evaluate the efficacy, safety and PK profile of GenSci140 in the treatment of ovarian cancer or other FRα-positive advanced solid tumors at different dose levels, and to select an appropriate RP2D (if applicable).

ELIGIBILITY:
Inclusion Criteria:

1. Those who are able to understand and willing to sign written Informed Consent Form.
2. Aged between 18 and 75 years (inclusive) when signing the ICF
3. Participants with advanced solid tumors
4. The participant agrees to provide fresh biopsy or archived tumor tissues for testing by the central laboratory.
5. At least one evaluable lesion in the dose-escalation part, and at least one measurable lesion in the dose-expansion part.
6. Eastern Cooperative Oncology Group performance status (ECOG PS) 0 or 1.
7. Life expectancy ≥ 3 months.
8. Adequate hematologic and organ function before the first dose of GenSci140.
9. All toxicities related to prior anti-tumor therapies must have resolved to Grade ≤ 1, with the following exceptions: alopecia, peripheral neurotoxicity (must have resolved to Grade ≤ 2).
10. For participants with congestive heart failure (CHF), it must be Grade ≤ 1 in severity and must have recovered completely prior to enrollment.
11. Normal QT interval on electrocardiogram (ECG) evaluation at screening
12. Participants who test negative for human immunodeficiency virus (HIV), hepatitis B virus (HBV), and hepatitis C virus (HCV).
13. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test result. WOCBP must agree to avoid pregnancy.
14. Men with female partners of childbearing potential must take appropriate precautions to avoid pregnancy of partner and use appropriate barrier contraceptives or abstinence

Exclusion Criteria:

1. Past history of cancers.
2. Symptomatic primary central nervous system (CNS) tumors, metastases, leptomeningeal carcinomatosis, or therapy naive spinal cord compression.
3. Use of an investigational medicinal product (IMP) or antitumor therapy (including chemotherapy, biologic therapy, immunotherapy) within 5 half-lives or 4 weeks before the first dose of GenSci140. Concomitant anti-tumor therapy is not permitted
4. Major surgery within 4 weeks prior to the first dose of GenSci140.
5. Radiotherapy for ≥ 20% of bone marrow or large area of radiotherapy within 4 weeks prior to the first dose of GenSci140. Or participants have not recovered from acute effects of radiotherapy to baseline prior to the first dose of GenSci140.
6. Clinically significant active cardiovascular disorder or history of myocardial infarction within 6 months prior to the first dose of GenSci140.
7. Uncontrolled active systemic bacterial, viral, or fungal infection or ongoing serious systemic disease, such as hypertension or diabetes, despite Best Supportive Care. Chronic disease screening is not required.
8. History of multiple sclerosis or other demyelinating diseases, Eaton-Lambert syndrome (paraneoplastic syndrome), alcoholic liver disease, history of internal haemorrhage or ischemic stroke within the past 6 months, haemorrhagic diathesis that are unsuitable for enrollment as assessed by the investigator.
9. Suspected treatment-related pneumonitis that was clinically diagnosed in the past and currently requires steroids or cannot be ruled out by imaging at screening.
10. Uncontrolled pleural effusion, pericardial effusion, or abdominal and pelvic fluid collection requiring drainage and/or diuretics within 14 days prior to the first dose of GenSci140.
11. Pregnant or lactating women.
12. Known hypersensitivity to prior monoclonal antibody therapy.
13. Patients who previously underwent allogeneic or autologous bone marrow transplantation.
14. Participants whom the investigator deems unsuitable for enrollment in this clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse event (AEs), and incidence of dose limiting toxicities（DLTs） | 3 weeks
  To determine the MTD (if any) of GenSci140 in participants with advanced solid tumors
maximal tolerance dose （MTD） | up to 3 months
  To determine the MTD (if any) of GenSci140 in participants with advanced solid tumors
recommended dose of expansion （RDE） | up to 3 months
  To determine the RDE of GenSci140 in participants with advanced solid tumors
objective response rate（ORR） | up to 5 months
  To evaluate the preliminary efficacy of GenSci140 in participants with advanced solid tumors
duration of response（DOR） | up to 5 months
  To evaluate the preliminary efficacy of GenSci140 in participants with advanced solid tumors
disease control rate（DCR） | up to 5 months
  To evaluate the preliminary efficacy of GenSci140 in participants with advanced solid tumors
Incidence and severity of adverse event (AEs) | up to 5 months
  To evaluate the safety and tolerability of GenSci140 at specific doses in participants with specific advanced solid tumors.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of China Medical University, Shenyang, Liaoning, China